CLINICAL TRIAL: NCT00071201
Title: A Multi-Center Phase 3, Open-Label, Parallel-Group Study to Evaluate the Efficacy, Safety and Pharmacokinetics of Adefovir Dipivoxil Liquid Suspension in Patients With Chronic Hepatitis B and Varying Degrees of Renal Impairment
Brief Title: Evaluate Efficacy, Safety and PK of Adefovir Dipivoxil Liquid Suspension in Patients With Chronic Hepatitis B
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-02-526
Record Dates: First submitted 2003-10-15; First posted 2003-10-17 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — adefovir dipivoxil; Suspensions

INTERVENTIONS:
Drug: Adefovir Dipivoxil for oral suspension, 2 mg/mL

SUMMARY:
This is a multi-center phase 3, open-label, parallel-group study designed to evaluate the efficacy, safety and pharmacokinetics of adefovir dipivoxil liquid suspension in patients with chronic hepatitis B and varying degrees of renal impairment.

DETAILED DESCRIPTION:
Approximately 48 patients with chronic hepatitis B will be enrolled into four groups representing varying degrees of renal function. Grouping will be achieved through estimation of creatinine clearance (CLcr) using the Cockcroft-Gault method of calculation at the time of screening:

Group 1: Mild (Clcr = greater than or equal to 50 to less than 80 mL/min)

Group 2: Moderate (Clcr = greater than or equal to 20 to less than 50 mL/min)

Group 3: Severe (Clcr = greater than or equal to 10 to less than 20 mL/min)

Group 4A-B: End stage renal disease (ESRD) including hemodialysis:

* Group 4A (Clcr = less than 10 mL/min)
* Group 4B (Patients undergoing hemodialysis)

At the baseline visit (day 0), blood and urine samples will be collected pre-dose (prior to 0 hour) after which patients will receive an oral dose of liquid adefovir dipivoxil according to the treatment guideline outlined in the protocol.

Pharmacokinetic parameters in plasma will be determined for the day 0 and week 12 visits for all patients and at the week 48 visit for group 1, 2, 3, and 4A patients. Pharmacokinetic parameters in urine will be determined for the day 0, week 12 and week 48 visits for group 1, 2, 3, and 4A patients.

At week 4, 8, 16, 20, 24, 28, 32, 36, 40, and 44 visits, pharmacokinetic assessments in plasma will be determined pre-dose (Ctrough levels) in groups 1, 2, 3, and 4A. For group 4B patients, pharmacokinetic assessments will be determined at weeks 4 and 8 prior to and upon completion of hemodialysis.

Evaluations of safety and efficacy will be conducted at 4 weekly intervals up to week 48 for groups 1, 2, 3, and 4A, and up to week 12 for group 4B. At these visits, patients will receive the next study medication allocation. Study medication administration will continue for up to a total of 48 weeks.

ELIGIBILITY:
INCLUSION CRITERIA:

* Male or female ages 18 through 65 years
* Able to give written informed consent and comply with the requirements of the study
* Females of childbearing potential must have a negative serum pregnancy test at screening and must use effective methods of contraception throughout the study.
* Positive serum HBV DNA equal to or greater than 100,000 copies/mL
* Patients with abnormal renal function, defined as a calculated creatinine clearance less than 80 mL/min, or end stage renal disease undergoing hemodialysis
* For non-hemodialysis patients, renal function must be "stable"
* ALT value equal to or greater than 1.2 to equal to or less than 15 times the upper limit of normal on at least two occasions, or histological evidence of necroinflammation and/or fibrosis
* Compensated liver disease with the following:

  * Prothrombin time equal to or less than to 1 second above normal range
  * Total bilirubin equal to or less than to 2.5 mg/dL or normal direct bilirubin
* No history of variceal bleeding or encephalopathy
* HIV, HCV, and HDV seronegative
* Adequate hematological function defined as:

  * Absolute neutrophil count equal to or greater than 750/mm3
  * Platelets equal to or greater than 50,000/mm3
  * Hemoglobin equal to or greater than 7.5 g/dL

EXCLUSION CRITERIA:

* Inability to comply with study requirements
* Lactating or pregnant females
* History or current manifestations of clinically significant cardiac, respiratory, endocrine (including diabetes mellitus), metabolic, gastrointestinal, dermatological, infectious, malignant, hematological, neurological, rheumatologic or psychiatric disorder, which is not related to the patient's renal insufficiency or deemed by the investigator to preclude suitability for pharmacokinetic assessment or interfere with patient treatment, assessment, or compliance with the protocol
* Received interferon within 6 months prior to study screening
* Bone marrow transplant recipients
* Renal transplant less than 6 months prior to study entry, or clinical evidence of rejection
* Patients expected to receive organ transplantation within 48 weeks
* Evidence of active liver disease due to other causes
* Patients taking chemotherapeutic agents within 2 months or expected to receive these agents during the study
* Previous participation in an investigational trial involving any investigational compound within 2 months, or within 5 half-lives of the study drug if sooner
* History of alcohol or drug abuse sufficient to hinder compliance with protocol
* Child-Pugh-Turcotte score over 9
* Evidence of hepatic mass suggestive of hepatocellular carcinoma
* History of malignancy other than basal cell carcinoma or treated cervical carcinoma in situ or cervical dysplasia
* The use of systemic drugs with potential activity against HBV for a period of more than 12 weeks in duration at any time
* The use of adefovir dipivoxil for a period of more than 12 weeks in duration at any time. Hemodialysis patients may be enrolled regardless of prior treatment duration with adefovir dipivoxil if treatment completed greater than or equal to 16 weeks before study.
* Hypersensitivity to nucleoside and/or nucleotide analogs
* Received hepatotoxic drugs within 2 months or plan to receive them
* Received nephrotoxic drugs or competitors of renal excretion within 2 months or plan to receive them, except for transplant patients
* Current use of other pivalic acid containing medications
* Patients undergoing continuous ambulatory peritoneal dialysis (CAPD)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48
Dates: Start 2003-06; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Gilead Sciences, Inc. 333 Lakeside Drive, Foster City, California, United States

REFERENCES:
- [Background] Hadziyannis SJ, Tassopoulos NC, Heathcote EJ, Chang TT, Kitis G, Rizzetto M, Marcellin P, Lim SG, Goodman Z, Wulfsohn MS, Xiong S, Fry J, Brosgart CL; Adefovir Dipivoxil 438 Study Group. Adefovir dipivoxil for the treatment of hepatitis B e antigen-negative chronic hepatitis B. N Engl J Med. 2003 Feb 27;348(9):800-7. doi: 10.1056/NEJMoa021812. PMID 12606734
- [Background] Marcellin P, Chang TT, Lim SG, Tong MJ, Sievert W, Shiffman ML, Jeffers L, Goodman Z, Wulfsohn MS, Xiong S, Fry J, Brosgart CL; Adefovir Dipivoxil 437 Study Group. Adefovir dipivoxil for the treatment of hepatitis B e antigen-positive chronic hepatitis B. N Engl J Med. 2003 Feb 27;348(9):808-16. doi: 10.1056/NEJMoa020681. PMID 12606735
- [Background] Westland CE, Yang H, Delaney WE 4th, Gibbs CS, Miller MD, Wulfsohn M, Fry J, Brosgart CL, Xiong S; 437 and 438 Study Teams. Week 48 resistance surveillance in two phase 3 clinical studies of adefovir dipivoxil for chronic hepatitis B. Hepatology. 2003 Jul;38(1):96-103. doi: 10.1053/jhep.2003.50288. PMID 12829991
- See also: Gilead's website — http://www.gilead.com
- See also: Study Results — http://www.gileadclinicaltrials.com/pdf/GS-02-526_synopsis.pdf